CLINICAL TRIAL: NCT04379635
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Compare the Efficacy and Safety of Neoadjuvant Treatment With Tislelizumab (BGB-A317, Anti-PD-1 Antibody) or Placebo Plus Platinum-Based Doublet Chemotherapy Followed By Adjuvant Tislelizumab or Placebo in Resectable Stage II or IIIA Non-Small Cell Lung Cancer
Brief Title: Comparing the Efficacy and Safety of a New Additional Treatment With Tislelizumab in Non-Small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BGB-A317-315; CTR20200821 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Cisplatin; Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy + Neoadjuvant/Adjuvant Tislelizumab (Experimental): Tislelizumab + cisplatin/carboplatin + paclitaxel or Pemetrexed Disodium
  Interventions: Drug: Tislelizumab; Drug: Cisplatin injection; Drug: Paclitaxel injection; Drug: Pemetrexed Disodium; Drug: Carboplatin
- Neoadjuvant chemotherapy + Neoadjuvant/Adjuvant Placebo (Placebo Comparator): Placebo + cisplatin/carboplatin + paclitaxel or Pemetrexed Disodium
  Interventions: Drug: Cisplatin injection; Drug: Paclitaxel injection; Drug: Pemetrexed Disodium; Drug: Placebos; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — administered via Intravenous (IV) injection
  Other Names: BGB-A317
  Arms: Neoadjuvant chemotherapy + Neoadjuvant/Adjuvant Tislelizumab
Drug: Cisplatin injection — administered via IV infusion
Drug: Paclitaxel injection — administered via IV infusion
Drug: Pemetrexed Disodium — administered via IV infusion
Drug: Placebos — Placebo to match tislelizumab IV infusion
  Arms: Neoadjuvant chemotherapy + Neoadjuvant/Adjuvant Placebo
Drug: Carboplatin — administered via IV infusion

SUMMARY:
The primary objective of this study is to evaluate and compare major pathological response(MPR) rate and event-free survival (EFS) in participants receiving tislelizumab plus platinum-based doublet chemotherapy as the new additional treatment followed by tislelizumab as adjuvant treatment versus participants receiving placebo plus platinum-based doublet chemotherapy as neoadjuvant treatment followed by placebo as adjuvant treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
2. Histologically confirmed Stage II or IIIA NSCLC
3. Measurable disease as assessed per RECIST v1.1
4. Confirm eligibility for an R0 resection with curative intent

Key Exclusion Criteria:

1. Any prior therapy for current lung cancer, including chemotherapy, or radiotherapy
2. Known Epidermal growth factor receptor (EGFR) mutation or Anaplastic Lymphoma Kinase (ALK) gene translocation
3. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days before randomization
4. Active autoimmune diseases or history of autoimmune diseases that may relapse
5. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) in Intent-to-Treat (ITT) analysis set | Up to 3 months following completion of neoadjuvant treatment
Event-free survival (EFS) in ITT analysis set as Assessed by the Blinded Independent Central Review (BICR) | Up to 5 years

SECONDARY OUTCOMES:
Overall survival (OS) in the ITT set | Up to 5 years
Pathological complete response (pCR) rate | Up to 5 years
Objective Response Rate (ORR) | Up to 5 years
Disease-Free Survival (DFS) in ITT analysis set | Up to 5 years
Event-free survival (EFS) Assessed by the Investigator | Up to 5 years
Number of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 5 years
Efficacy and Safety as Assessed by Health-related quality of life (HRQoL) Questionnaire | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (44):
- China (44):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences (Ningbo No Hospital), Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Derived] Wang C, Wang W, Liu H, Chen Q, Chen C, Liu L, Zhang P, Zhao G, Yang F, Han G, Yu B, Yang Y, Chen H, Jiang J, Tan L, Xu S, Mao N, Hu J, Zhang L, Zhang Z, Yao B, Wang S, Leaw S, Naicker K, Zheng W, Yu C, Yue D; RATIONALE-315 investigators. Perioperative tislelizumab plus neoadjuvant chemotherapy for patients with resectable non-small-cell lung cancer: final analysis of the randomized RATIONALE-315 trial. Ann Oncol. 2025 Dec 2:S0923-7534(25)06287-8. doi: 10.1016/j.annonc.2025.11.017. Online ahead of print. PMID 41344593
- [Derived] Yue D, Wang W, Liu H, Chen Q, Chen C, Liu L, Zhang P, Zhao G, Yang F, Han G, Cheng Y, Yu B, Yang Y, Chen H, Jiang J, Tan L, Xu S, Mao N, Hu J, Zhang L, Yao B, Wang S, Wang RH, Zheng W, Wang C; RATIONALE-315 investigators. Perioperative tislelizumab plus neoadjuvant chemotherapy for patients with resectable non-small-cell lung cancer (RATIONALE-315): an interim analysis of a randomised clinical trial. Lancet Respir Med. 2025 Feb;13(2):119-129. doi: 10.1016/S2213-2600(24)00269-8. Epub 2024 Nov 21. PMID 39581197